CLINICAL TRIAL: NCT05696574
Title: Comparative Study Between Oral and Vaginal Misoprostol for Induction of Labor in Nulliparous Pregnant Women at or Beyond Completed 41 Weeks
Brief Title: Oral and Vaginal Misoprostol for Induction of Labor in Nulliparous Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elsayed Fekry Elsayed Omran, Obstetrics and Gynecology Resident, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-35-2022
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Misoprostol; Labor; Nulliparous; Pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Misoprostol group (Experimental): Women in this group will include 40 pregnant women who will be offered misoprostol (placed in the post-fornix of the vagina) in a dose of 25µg to be repeated every 6 hours if no response is achieved with a maximum of 4 doses.
  Interventions: Drug: Vaginal Misoprostol
- Oral Misoprostol group (Experimental): Women in this group will include 40 pregnant women who will be offered oral misoprostol in a dose of 25µg to be repeated every 6 hours if no response is achieved with a maximum of 4 doses.
  Interventions: Drug: Oral Misoprostol

INTERVENTIONS:
Drug: Vaginal Misoprostol — Women in this group will include 40 pregnant women who will be offered misoprostol (placed in the post-fornix of the vagina) in a dose of 25µg to be repeated every 6 hours if no response is achieved with a maximum of 4 doses.
  Arms: Vaginal Misoprostol group
Drug: Oral Misoprostol — Women in this group will include 40 pregnant women who will be offered oral misoprostol in a dose of 25µg to be repeated every 6 hours if no response is achieved with a maximum of 4 doses.
  Arms: Oral Misoprostol group

SUMMARY:
The aim of this study is to compare the efficacy and the safety of vaginal misoprostol with oral misoprostol for induction of labor in nulliparous pregnant women at or beyond completed 41 weeks.

DETAILED DESCRIPTION:
Induction of labor is carried out for maternal and fetal indications and one of the most common indications is prolonged pregnancy.

Recent studies have suggested that by continuing pregnancy beyond 41 weeks, there is statistically significantly higher perinatal morbidity and mortality as well as an increased risk to the mother. Thus, there is a growing body of evidence suggesting the elective induction of labor at 41 weeks of gestation instead of expectant management.

Misoprostol, a prostaglandin E1 analog, is indicated for protection against gastric ulcers, but when administered prenatally it causes uterine contractions. Research exploiting this adverse effect has shown misoprostol to be superior to conventional methods for induction, resulting in shorter induction-to-delivery intervals, without any increase in adverse outcomes. It has the advantage of being cheap, stable at room temperature, and easy to be administered by various routes i.e., vaginal, oral, sublingual, or rectal.

The differential outcomes of oral versus vaginal misoprostol may be secondary to different pharmacokinetics for oral compared with vaginal misoprostol. Oral misoprostol undergoes rapid absorption from the gastrointestinal tract and rapid and extensive de-esterification during first-pass metabolism to an active metabolite, misoprostol, peaking at 15 minutes with a half-life of 20-40 minutes. Misoprostol then undergoes early rapid elimination over 120 minutes, followed by slow elimination thereafter. The medication rapidly makes its way to the myometrium. ln contrast, after vaginal misoprostol administration, plasma concentration gradually increase, reaching a maximum level after 70-80 minutes before slowly being eliminated with plasma levels still detectable 6 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age: 18-40.
2. Nullipara: a woman who has never completed a pregnancy beyond 20 weeks gestation. She may not have been pregnant or may have had a spontaneous or elective abortion(s) or an ectopic pregnancy.
3. Single living pregnancy.
4. Gestational age: at or beyond completed 41 weeks (confirmed by a reliable date for the last menstrual period, regular cycle, or/and 1st trimesteric ultrasound scan).
5. Cephalic presentation.
6. Bishop score of 6 or less.
7. Reactive fetal non-stress test (NST).

Exclusion Criteria:

1. Any maternal chronic diseases or pregnancy-induced medical disorders.
2. Fetal anomalies.
3. Fetal macrosomia (>4 Kg).
4. Intrauterine Growth Restriction (IUGR) (EFW below the 10th percentile for gestational age).
5. Rupture of membranes or oligohydramnios (AFI < the fifth percentile).
6. Previous uterine scar.
7. Regular uterine contractions.
8. Any contraindication to vaginal delivery e.g., placenta previa (complete or partial covering of the internal os of the cervix with the placenta).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Nulliparous pregnant women who are candidates for induction of labor at or beyond completed 41 weeks
Enrollment: 80 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Onset of active stage of labor | 24 hours postoperatively
  Duration to onset of active stage of labor

SECONDARY OUTCOMES:
Cesarean section rate in each group | Within 24 hours from drug induction
  Cesarean section rate will be recorded
Doses given | Intraoperativley
  Number of durg doses given will be recored
Augmentation need | Intraoperatively
  Number of participants need for labor augmentation with oxytocin and/or amniotomy will be evaluated
Complications | 48 hours Postoperatively
  Any complications will be recorded

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study